CLINICAL TRIAL: NCT01218516
Title: A Randomized, Double-Blind, Placebo-Controlled, Study of the Safety and Efficacy of Farletuzumab in Combination With a Platinum-Containing Doublet in Chemotherapy-Naive Subjects With Stage IV Adenocarcinoma of the Lung (FLAIR)
Brief Title: A Safety and Efficacy Study of Farletuzumab in Participants With Adenocarcinoma of the Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MORAb-003-009; 2010-022229-13 (EudraCT Number)
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2018-03

CONDITIONS: Adenocarcinoma of the Lung
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — farletuzumab; Carboplatin; Paclitaxel; Pemetrexed; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Farletuzumab plus Chemotherapy (Active Comparator): During Combination Therapy, farletuzumab will be given with a protocol-approved platinum doublet (either carboplatin/paclitaxel, carboplatin/pemetrexed, or cisplatin/pemetrexed) for at least 4, but not more than 6, cycles. Participants who experience clinical benefit from the Combination Therapy will enter the Monotherapy Phase and receive farletuzumab as monotherapy until disease progression.
  Interventions: Biological: Farletuzumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Cisplatin
- Placebo plus Chemotherapy (Placebo Comparator): During Combination Therapy, placebo will be given with a protocol-approved platinum doublet (either carboplatin/paclitaxel, carboplatin/pemetrexed, or cisplatin/pemetrexed) for at least 4, but not more than 6 cycles. Participants who experience clinical benefit from the Combination Therapy will enter the Monotherapy Phase and receive placebo as monotherapy until disease progression.
  Interventions: Other: Placebo; Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Biological: Farletuzumab — Combination Therapy: Farletuzumab 7.5 mg/kg will be administered intravenously on Cycle 1, Week 1 and Cycle 1, Week 2 (loading dose). Beginning on Cycle 2, Week 1, farletuzumab (7.5 mg/kg) will be administered intravenously on Week 1 of all additional cycles.
  Monotherapy: Farletuzumab 7.5 mg/kg will be administered intravenously on Week 1 of every 3-week cycle until disease progression.
  Other Names: MORAb-003
  Arms: Farletuzumab plus Chemotherapy
Other: Placebo — Combination Therapy: Placebo will be administered intravenously on Cycle 1, Week 1 and Cycle 1, Week 2 (loading dose). Beginning on Cycle 2, Week 1, placebo will be administered IV on Week 1 of all additional cycles.
  Monotherapy: Placebo will be administered intravenously on Week 1 of every 3-week cycle until disease progression.
  Arms: Placebo plus Chemotherapy
Drug: Carboplatin — Carboplatin will be administered intravenously to achieve area under the serum concentration-time curve of 5 to 6 mg/mL^min [AUC5-6].
Drug: Paclitaxel — Paclitaxel 200 mg/m^2 will be administered intravenously.
Drug: Pemetrexed — Pemetrexed 500 mg/m^2 will be administered intravenously.
Drug: Cisplatin — Cisplatin 75 mg/m^2 will be administered intravenously.

SUMMARY:
The primary objective of this study is to compare the effect of farletuzumab versus placebo in combination with either a platinum agent (carboplatin) with paclitaxel or a platinum agent (carboplatin or cisplatin) with pemetrexed followed by farletuzumab or placebo on investigator-assessed progression free survival (PFS) as determined by Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 or definitive clinical disease progression (eg, new occurrence of positive fluid cytology) in chemotherapy naive participants with folate receptoralpha (FRA)-expressing Stage IV adenocarcinoma of the lung.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the lung classified as stage IV
* Confirmed folate receptor-alpha (FRA) expression by immunohistochemistry (IHC)
* Measurable disease with at least one unidimensionally measurable lesion according to RECIST criteria version 1.1 by computed tomography (CT) or magnetic resonance imaging (MRI) scans (CT or MRI scans must have been performed within 30 days prior to the first dose of farletuzumab or placebo)
* Must have received no prior chemotherapy, radiation therapy or surgery with curative intent for adenocarcinoma of the lung

Exclusion Criteria:

* Participants who have had previous chemotherapy for adenocarcinoma of the lung
* Prior surgery with curative intent for adenocarcinoma of the lung
* Prior radiotherapy for adenocarcinoma of the lung. (Prior treatment with local radiotherapy for symptom control [i.e., palliative radiation with non-curative intent] is permitted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-06-27 (Actual); Primary Completion 2012-12-15 (Actual); Study Completion 2013-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (93):
- United States (54):
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - Arizona Center for Hematology Oncology, Glendale, Arizona
  - Providence Health System, Beverly Hills, California
  - Cancer Care Associates of Fresno Medical Group, Inc., Fresno, California
  - Medical Oncology Hematology, Gilroy, California
  - California Cancer Care, Inc., Greenbrae, California
  - Moores University of California San Diego Cancer Center, La Jolla, California
  - Wilshire Medical Oncology Group, La Verne, California
  - Glendale Adventist Medical Center, Los Angeles, California
  - Clinical Trials and Research Associates, Inc., Montebello, California
  - North Country Oncology-Hematology, Oceanside, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Central Coast Medical Oncology, Santa Maria, California
  - Rocky Mountain Cancer Centers, LLP, Denver, Colorado
  - Hematology Oncology Associates, P.C., Stamford, Connecticut
  - Center for Hematology-Oncology, Boca Raton, Florida
  - Medical Specialists of the Palm Beaches, Deerfield Beach, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Cancer Care of North Florida, Lake City, Florida
  - Florida Cancer Institute-New Hope, New Port Richey, Florida
  - Ocala Oncology Center, PL, Ocala, Florida
  - MD Anderson Cancer Center-Orlando, Orlando, Florida
  - University Hematology Oncology, Inc., Centralia, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - The Community Hospital, Munster, Indiana
  - Kentucky Cancer Center, Hazard, Kentucky
  - Baptist Health System, Inc., Lexington, Kentucky
  - Christus Saint Frances, Cabrini Hospital, Cabrini Cancer Center, Alexandria, Louisiana
  - Hematology and Oncology Specialists, LLC, Metairie, Louisiana
  - National Cancer Institute, Bethesda, Maryland
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Queens Hospital Center, Jamaica, New York
  - Syracuse Veterns Affairs Medical Center, Syracuse, New York
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - St. Luke's Cancer Center Associates, Bethlehem, Pennsylvania
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Texas Oncology - Bedford, Bedford, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Houston Cancer Institute, Houston, Texas
  - Texas Oncology - Plano East, Plano, Texas
  - Northwest Cancer Center, Sugar Land, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Texas Oncology - Waco, Waco, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Delta Hematology Oncology Associates, PC, Portsmouth, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Rockwood Cancer Treatment Center, Spokane, Washington
  - Medical Oncology Associates, PS, Spokane, Washington
  - Cancer Team Bellin Health, Green Bay, Wisconsin
- Australia (12):
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Southern Medical Day Oncology Care Centre, Wollongong, New South Wales
  - Royal Brisbane and Women's Hospital, Dept. of Medical Oncology, Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Cancer Centre, Adelaide, South Australia
  - Flinders Medical Centre, Dept. of Oncology, Bedford Park, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Frankston Hospital, Oncology Day Unit, Frankston, Victoria
  - Epworth Healthcare, Richmond, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- Canada (4):
  - Royal Victoria Hospital, Barrie, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Germany (8):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinik Löwenstein gGmbH, Löwenstein, Baden-Wurttemberg
  - Asklepios Fachkliniken München-Gauting, Gauting, Bavaria
  - Krankenhaus Nordwest GmbH, Frankfurt am Main, Hesse
  - Johannes-Wesling-Klinikum Minden, Minden, North Rhine-Westphalia
  - Städtisches Krankenhaus Martha-Maria Halle Dölau gGmbH, Halle, Saxony-Anhalt
  - HELIOS Klinikum Emil von Behring, Berlin
  - Asklepios Klinik Harburg, Hamburg
- Italy (4):
  - Ospedale Unico Versilia, Lido di Camaiore, Lucca
  - Azienda Ospedaliero-Univesitaria "San Luigi Gonzaga", Orbassano, Torino
  - Istituto Nazionale per la Ricerca sul Cancro, Genova
  - A.O. Seconda Università degli Studi di Napoli, Napoli
- Poland (3):
  - Wojewódzki Szpital Zespolony im. L. Rydygiera w Toruniu Szpital Dzieciecy, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Onkologii - Instytut im. M. Sklodowskiej-Curie w Warszawie, Warsaw, Masovian Voivodeship
  - Specjalistyczny Szpital im. Alfreda Sokolowskiego, Szczecin, West Pomeranian Voivodeship
- Russia (3):
  - Republican Clinical Oncologic Dispensary of Ministry of health of Republic Tatarstan, Kazan', Tatarstan Republic
  - Cancer Research Center n.a. N.N. Blokhin, Moscow
  - City Oncology Hospital # 62, Moscow
- Spain (5):
  - Hospital Regional Carlos Haya, Málaga, Malaga
  - Hospital General Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Germans Trías i Pujol, Barcelona
  - Fundación Jiménez Díaz, Madrid

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All screening procedures were completed within 30 days prior to and including the Cycle 1 Day 1 Visit.
Groups:
- Combination Therapy: Placebo + Chemotherapy: During Combination Therapy, placebo was given with a protocol-approved platinum doublet (either carboplatin/paclitaxel, carboplatin/pemetrexed, or cisplatin/pemetrexed) for at least 4, but not more than 6, cycles. Duration of each cycle=3 weeks.
- Combination Therapy: Farletuzumab + Chemotherapy: During Combination Therapy, farletuzumab was given with a protocol-approved platinum doublet (either carboplatin/paclitaxel, carboplatin/pemetrexed, or cisplatin/pemetrexed) for at least 4, but not more than 6 cycles. Duration of each cycle=3 weeks.
- Monotherapy: Placebo: Following at least 4 cycles, but not more than 6 cycles of combination therapy, participants who experienced clinical benefit from the Combination Therapy (Placebo + Chemotherapy) entered the Monotherapy phase and received placebo as monotherapy until disease progression. Duration of each cycle=3 weeks.
- Monotherapy: Farletuzumab: Following at least 4 cycles, but not more than 6 cycles of combination therapy, participants who experienced clinical benefit from the Combination Therapy (Farletuzumab + Chemotherapy) entered the Monotherapy phase and received farletuzumab as monotherapy until disease progression. Duration of each cycle=3 weeks.
Period: Combination Therapy (up to 4.5 Months)
Arm/Group | Combination Therapy: Placebo + Chemotherapy | Combination Therapy: Farletuzumab + Chemotherapy | Monotherapy: Placebo | Monotherapy: Farletuzumab
Started | 67 | 63 | 0 | 0
Completed | 38 | 28 | 0 | 0
Not Completed | 29 | 35 | 0 | 0
Not completed — Death | 2 | 1 | 0 | 0
Not completed — Delay in TA Administration of >=28 days | 0 | 3 | 0 | 0
Not completed — Physician Decision | 2 | 2 | 0 | 0
Not completed — Chemotherapy Discontinued | 2 | 0 | 0 | 0
Not completed — Progressive Disease (PD) by RECIST v 1.1 | 17 | 15 | 0 | 0
Not completed — Randomized but Not Treated | 0 | 1 | 0 | 0
Not completed — Withdrew Consent | 0 | 1 | 0 | 0
Not completed — Deterioration of Performance Status | 0 | 3 | 0 | 0
Not completed — Other | 3 | 4 | 0 | 0
Not completed — Toxicity to TA | 0 | 1 | 0 | 0
Not completed — Participant Discontinued Treatment | 2 | 3 | 0 | 0
Not completed — Treatment With Items Outside Protocol | 1 | 1 | 0 | 0
Period: Monotherapy (up to 23.5 Months)
Arm/Group | Combination Therapy: Placebo + Chemotherapy | Combination Therapy: Farletuzumab + Chemotherapy | Monotherapy: Placebo | Monotherapy: Farletuzumab
Started | 0 (This phase ended once all participants finished.) | 0 (This phase ended once all participants finished.) | 38 (Only eligible participants entered this phase of the study.) | 28 (Only eligible participants entered this phase of the study.)
Safety Analysis Set | 0 | 0 | 35 | 31 (Three participants were randomized to placebo but actually received Farletuzumab.)
Completed | 0 | 0 | 38 | 28
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Therapy: Placebo + Chemotherapy | Combination Therapy: Farletuzumab + Chemotherapy | Total
Number analyzed (Participants) | 67 | 63 | 130
Age, Continuous [Median (Full Range); unit: Years] | 61.0 [46 to 79] | 60.0 [38 to 80] | 61.0 [38 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 41 | 34 | 75

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of the first observation of investigator-assessed (radiology review) progression based on Response Evaluation Criteria In Solid Tumors (RECIST) v.1.1 or other protocol-approved measures of disease progression (e.g., new occurrence of positive fluid cytology, newly diagnosed evidence of disease progression from histologic samples, PET-positive metastases, or new bone or brain metastases), or date of death, whatever the cause. Disease progression as assessed by the investigator per RECIST v1.0 was defined as at least a 20% increase in sum of longest diameters (RECIST definition) compared to baseline (or lowest sum while on study if less than baseline), or any new lesions (measurable or nonmeasurable).
Time Frame: From date of first administration of study drug up to 6 month follow-up from randomization of the last participant, i.e., cut-off date 15 Dec 2012 for primary analysis and cut-off date of 1 Nov 2013 or up to approximately 28 months for final analysis
Population: The ITT population included all randomized participants who received at least 1 dose of test article (placebo or farletuzumab), with treatment assignments designated according to actual study treatment received. This was the primary analysis population for evaluating treatment administration, tolerability, and safety.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy: Placebo + Chemotherapy | Combination Therapy: Farletuzumab + Chemotherapy
Number analyzed (Participants) | 67 | 63
Months
  Per Primary Analysis Cut-Off Date | 5.8 [5.0 to 6.8] | 4.7 [4.2 to 5.6]
  Per Final Analysis Cut-Off Date | 5.9 [5.0 to 7.0] | 4.7 [4.2 to 5.6]
Statistical Analysis 1: Comparison: Combination Therapy: Placebo + Chemotherapy vs Combination Therapy: Farletuzumab + Chemotherapy; Test type: Superiority or Other; p = 0.3519, Log Rank — Per Primary Analysis Cut-Off Date; Hazard Ratio (HR) = 1.23, 80% CI 2-sided [0.92 to 1.63]
Statistical Analysis 2: Comparison: Combination Therapy: Placebo + Chemotherapy vs Combination Therapy: Farletuzumab + Chemotherapy; Test type: Superiority or Other; p = 0.1555, Log Rank — Per Final Analysis Cut-Off Date; Hazard Ratio (HR) = 1.34, 80% CI 2-sided [1.03 to 1.74]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR, defined as the percentage of participants who had best overall response (BOR) of complete response (CR) or partial response (PR) as determined by investigator's radiologic assessments using RECIST 1.1 for target lesions and assessed by Magnetic resonance imaging (MRI) and computerized tomography (CT) scan (for double blind treatment period i.e. Randomization Phase). CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR = CR + PR.
Time Frame: From Day 1 until documented radiographic progression, other protocol-approved measures of disease progression, withdrawal by participant, death due to any cause, or cut-off date of 1 Nov 2013, i.e., up to approximately 28 months for final analysis
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Combination Therapy: Placebo + Chemotherapy | Combination Therapy: Farletuzumab + Chemotherapy
Number analyzed (Participants) | 67 | 63
Percentage of participants | 37.3 | 41.3

3. Secondary Outcome: Duration of Response (DR)
Description: DR was derived for those participants with objective evidence of CR or PR. DR was defined as the time (in months) from first documentation of objective response (CR or PR) to the first documentation of disease progression (ie, objective tumor progression as assessed by investigator's radiology review or other protocol-approved measures of disease progression) or death due to any cause. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the first documentation of objective response (CR or PR) to the first documentation of disease progression, death due to any cause, or cut-off date of 1 Nov 2013, i.e., up to approximately 28 months for final analysis
Population: Tumor Response (TR) Evaluable Analysis Set (responders only) included all participants who received at least 1 dose of test article and who had a baseline assessment and at least 1 on-treatment assessment performed, sufficient to assess the endpoint of interest. The TR Evaluable Analysis Set was used for all RECIST assessments of tumor response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy: Placebo + Chemotherapy | Combination Therapy: Farletuzumab + Chemotherapy
Number analyzed (Participants) | 25 | 25
Months | 6.7 [4.1 to 9.4] | 4.1 [3.0 to 7.0]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in months) from the date of randomization to the date of death, regardless of cause.
Time Frame: From the date of randomization to the date of death due to any cause or up to cut-off date of 1 Nov 2013 (up to approximately 28 months) for final analysis
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination Therapy: Placebo + Chemotherapy | Combination Therapy: Farletuzumab + Chemotherapy
Number analyzed (Participants) | 67 | 63
Months | 10.5 [8.3 to 14.0] | 14.1 [9.5 to 18.6]

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered with an investigational product. A serious adverse event (SAE) was defined as any untoward medical occurrence that at any dose; resulted in death, was life-threatening (i.e., the participant was at a risk of death at the time of the event; this did not include an event that hypothetically might have caused death if it had been more severe), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, or was a congenital abnormality/birth defect. In this study, TEAEs (defined as an AE that started/increased in severity on/after the first dose of study medication up to 30 days after the final dose of study medication) were assessed.
Time Frame: For each participant, from the first dose till 30 days after the last dose or cut-off date of 1 Nov 2013, i.e., up to approximately 28 months for final analysis
Population: The safety analysis set (SAS) included randomized participants who received at least 1 dose of test article, with treatment assignments designated according to actual study treatment received. This was the primary analysis population for evaluating treatment administration, tolerability, and safety.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy: Placebo + Chemotherapy | Combination Therapy: Farletuzumab + Chemotherapy | Monotherapy: Placebo | Monotherapy: Farletuzumab
Number analyzed (Participants) | 65 | 64 | 35 | 31
Participants
  TEAEs | 60 | 63 | 30 | 25
  Treatment emergent SAEs | 27 | 27 | 6 | 7

ADVERSE EVENTS:
Time Frame: For each participant, from the first dose till 30 days after the last dose or cut-off date of 1 Nov 2013, i.e., up to approximately 28 months for final analysis
Description: TEAEs, defined as an AE that started/increased in severity on/after the first dose of study drug up to 30 days after final dose of study drug. Per the study Statistical Analysis Plan, the TEAEs presented include serious and non-serious TEAEs. Additionally, serious TEAEs are presented separately.
Arm/Group | Combination Therapy: Placebo + Chemotherapy | Combination Therapy: Farletuzumab + Chemotherapy | Monotherapy: Placebo | Monotherapy: Farletuzumab
All-Cause Mortality (participants affected / at risk) | 46/65 | 39/64 | 1/35 | 0/31
Serious Adverse Events (participants affected / at risk) | 27/65 | 27/64 | 6/35 | 7/31
Other Adverse Events (participants affected / at risk) | 60/65 | 63/64 | 30/35 | 25/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy: Placebo + Chemotherapy (N=65) | Combination Therapy: Farletuzumab + Chemotherapy (N=64) | Monotherapy: Placebo (N=35) | Monotherapy: Farletuzumab (N=31)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy: Placebo + Chemotherapy (N=65) | Combination Therapy: Farletuzumab + Chemotherapy (N=64) | Monotherapy: Placebo (N=35) | Monotherapy: Farletuzumab (N=31)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Asthenia (General disorders) | 12 (13) | 22 (32) | 3 (3) | 2 (2)
Fatigue (General disorders) | 29 (48) | 24 (29) | 3 (4) | 1 (1)
Pyrexia (General disorders) | 6 (8) | 9 (15) | 1 (1) | 2 (3)
Mucosal inflammation (General disorders) | 9 (15) | 7 (7) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 5 (5) | 6 (8) | 3 (3) | 1 (2)
Chills (General disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 5 (6) | 6 (6) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (4) | 7 (7) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 4 (4) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 20 (24) | 24 (27) | 4 (5) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 10 (18) | 22 (34) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (11) | 8 (9) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (6) | 4 (6) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 12 (15) | 6 (6) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 9 (14) | 4 (4) | 6 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4) | 0 (0) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 6 (6) | 8 (10) | 0 (0) | 2 (4)
Headache (Nervous system disorders) | 1 (1) | 3 (4) | 1 (1) | 5 (5)
Paraesthesia (Nervous system disorders) | 8 (9) | 6 (7) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 5 (5) | 3 (3) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 6 (6) | 3 (3) | 1 (1) | 1 (1)
Polyneuropathy (Nervous system disorders) | 3 (3) | 4 (5) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 5 (11) | 3 (4) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 30 (48) | 29 (43) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 18 (26) | 20 (27) | 3 (6) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 16 (22) | 18 (21) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 16 (33) | 16 (25) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 7 (11) | 6 (8) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 4 (5) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (2) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 8 (9) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (7) | 4 (4) | 1 (2) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 9 (11) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (11) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 7 (8) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 5 (8) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 3 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 14 (21) | 17 (19) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 8 (10) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (6) | 7 (8) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (6) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (7) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 3 (3) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site urticaria (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Infusion site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral cyst (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paresis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Capillaritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Abdominal Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes dermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitic Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Respiratory tract infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (5) | 3 (3) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (4) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
C-Reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Weight increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (2)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 2 (3) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Renal fusion anomaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases To central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes